Planning for the Care You Want: A Counseling Intervention in the Outpatient Setting

PI: Ramona Rhodes, MD

UTSW IRB # 042016-050

Script for Obtaining Verbal Consent for Participation 9/8/2017

## **Recruitment Call Script**

This is [name of research staff] calling from UT Southwestern Medical Center. May I speak with [patient's name]?

Good [morning/afternoon/evening]. I'm calling to follow up on a letter you may have received within the last few days from Parkland and UT Southwestern inviting you to participate in a research study survey. Do you recall receiving that letter? [If patient has not received the letter, offer to read it to them or resend it. Then proceed with the call.]

I'd like to tell you a little about the survey and answer any questions you may have. Is this a good time to talk? [If so, proceed. Otherwise, arrange a time to call back.]

This survey is being done by Dr. Ramona Rhodes, an African American doctor at Parkland, who's interested in helping African American patients of Parkland Hospital better understand their options for care. We're inviting African Americans of the oncology clinic to participate by completing the survey over the phone. About 60 patients will participate in this study. The survey takes about 20 minutes. The questions are quite personal and some of them might make you uncomfortable. You can choose not to answer a question, take a break, or stop participation at any time. After completing the survey, you'll receive a \$10 gift card as a thank you for your time. There are no tests or procedures other than taking the survey.

Some patients who take the survey will be called by someone from the study team and invited to watch a short educational video at their next appointment. The video explains different options for planning for the care you want. Not everyone will be asked to watch the video—that's part of the design of the study. I don't know if you'll be contacted to watch the video or not. If so, you would be offered an additional \$20 gift card for meeting with the staff person and watching the video. After watching the video, the staff person can answer questions you might have. In addition, she'll follow up by phone during the next week to see if any questions come up about the topic and to offer help with referrals, if you. You do not have to agree to meet the staff person to watch the video, although we hope you will want to. We will not ask you to do anything beyond meeting the staff person and watching the video. We hope you would find the video enjoyable, though there's the slight risk some of the topics might make you feel uncomfortable.

If you do this first survey, we will call you again in one month, three months, and six months to invite you to do another short survey on the phone. These surveys take about 15 minutes. And like the first survey, you will receive a \$10 gift card as a thank you for your time after each one. You can choose to stop participating at any time. Again, you do not have to agree to participate in these surveys, but we hope you will want to.

If you have a friend or family member who is involved in your care or goes to your appointments with you, we're inviting them to take the survey as well. They, too, would receive a gift card for each survey they complete.

While participation in this study may not benefit you directly, we hope that responses to these surveys will help us find better ways to explain advance care planning to African American patients. If you decide to participate, the study doctor will look at your medical record to collect some information about your health. Although we take every precaution to make sure your information stays completely private, there's always the slight risk of loss of confidentiality. No reports or publications will use your name or other information that could identify you. Your survey responses will remain anonymous. If you have any questions or concerns, you can call Dr. Rhodes or myself at the phone number listed in the letter you received. That number is 214-648-8559.

Does this sound like something you might like to do?

[If the patient agrees . . .]

Do you have a friend or family member is your caregiver who might like to participate? [If yes...] Are they there with you now? [If yes...] May I speak with them? I'll tell them about the survey and see if it's something they'd like to do, then arrange a time to call them and do it.

[After the survey, verify address for sending gift card and best phone number for follow up. Then . . .]

As I said, someone from the study team may call you to arrange to meet you at your next appointment and show you the video. If they call, we hope you'll say yes. Do you have any questions for me? You can always call the study phone number and leave a message for someone to call you back.

Thank you very much.